CLINICAL TRIAL: NCT06506071
Title: Characterization of Acute Myocardial Damage With Spectral Computed Tomography. CADAMI-SPECTRAL.
Brief Title: Characterization of Acute Myocardial Damage With Spectral Computed Tomography. (CADAMI-SPECTRAL)
Acronym: CADAMI
Status: Recruiting | Type: Observational
Sponsor: Salamanca University Hospital (Other)
Collaborators: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Candelas Pérez del Villar, Principal investigator, Salamanca University Hospital
Other Study IDs: CADAMI-SPECTRAL
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Myocarditis; Acute or Subacute; Takotsubo Cardiomyopathy; Infarction, Myocardial; Myocardial Injury
MeSH Terms: conditions — Myocarditis; Takotsubo Cardiomyopathy; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Case: Myocardial tissue characterisation using spectral technology and Cardiac Magnetic Resonance (CMR) imaging.
  Interventions: Diagnostic Test: Spectral CT
- Controls: Myocardial tissue characterisation using spectral technology and CMR imaging.
  Interventions: Diagnostic Test: Spectral CT

INTERVENTIONS:
Diagnostic Test: Spectral CT — Myocardial tissue characterization with Spectral CT

SUMMARY:
Clinical management of patients with chest pain and elevation of biomarkers of myocardial injury require an accurate diagnosis. Until now, cardiac magnetic resonance imaging (cMRI) is the gold standard for the diagnosis among myocarditis, stress cardiomyopathy, or inapparent ischemic damage. The development of spectral CT has opened up the possibility of characterizing the coronary anatomy and the myocardium in a single procedure. Our aim is to assess the diagnostic ability of differential patterns in first- pass perfusion and delayed iodine enhancement obtained by spectral CT in patients with acute myocardial injury. This study is designed as a prospective multicenter observational study with diagnostic intervention in 150 patients admitted with clinical indication of a cMRI due to suspicion of myocardial infarction with normal coronary arteries (MINOCA), myocarditis or stress cardiomyopathy who will undergo a CT study with double detector technology in two reference centers. A control group (n=150) with an indication for cardiac CT for another cause without coronary or structural heart disease will be included. The iodine maps obtained by spectral CT will be compared with the findings obtained with cMRI, both with conventional techniques and with artificial intelligence algorithms (deep learning). A year follow-up of the cohort will be carried out to assess whether the findings derived from the CT in this group of patients provide prognostic information

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year.
* Hospital admission due to chest pain and acute myocardial injury.
* Clinical indication for cardiac MRI (CMR) due to suspected acute myocardial infarction with coronary angiography showing no significant lesions (<50%) (MINOCA), acute myocarditis, or stress-induced cardiomyopathy.
* Signed informed consent.

Exclusion Criteria:

* Contraindications to undergo cardiac MRI and CT with administration of gadolinium and/or iodine-based contrast, respectively.
* Pre-existing cardiomyopathy.
* Pre-existing chronic ischemic heart disease.
* Invasive coronary angiography showing coronary lesions ≥50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted with a suspected diagnosis of acute myocardial injury or subjects with a clinical indication for cardiac CT (CCT) for other reasons without myocardial injury or previous structural heart disease, with ≤1 cardiovascular risk factor, left ventricular ejection fraction > 55%, and absence of significant valvular disease (grade < III), with a similar age and sex distribution to cases with a clinical indication for CCT for other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between volume of myocardium with abnormal perfusion (measured using spectral iodine density images) and percentage of myocardium with late gadolinium enhacement -LGE- (measured by CMR). | 2 years
  To describe the differential alterations in first-pass and late iodine-enhanced images using spectral CT in patients diagnosed with MINOCA, myocarditis, and stress-induced cardiomyopathy, and comparing them with findings obtained by cardiac MRI.

SECONDARY OUTCOMES:
Characterize acute myocardial injury using spectral images obtained after the administration of iodine-based contrast in patients with MINOCA, acute myocarditis, and stress-induced cardiomyopathy, as well as in control subjects. | 2 years
  Characterize acute myocardial injury using spectral images obtained both in the early (first-pass) phase and in the late gadolinium-enhanced phase after the administration of iodine-based contrast in patients with MINOCA, acute myocarditis, and stress-induced cardiomyopathy, as well as in control subjects.
To describe the type of perfusion abnormality (hyperemia o perfusion deficit) which correlates with ischaemic and inflammatory,no ischemic myocardial injuries. | 2 years
  Assess whether spectral CT allows differentiation between the different etiologies of myocardial injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Asistencial Universitario de Salamanca. Instituto de Investigación Biomédica de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Townsend N, Kazakiewicz D, Lucy Wright F, Timmis A, Huculeci R, Torbica A, Gale CP, Achenbach S, Weidinger F, Vardas P. Epidemiology of cardiovascular disease in Europe. Nat Rev Cardiol. 2022 Feb;19(2):133-143. doi: 10.1038/s41569-021-00607-3. Epub 2021 Sep 8. PMID 34497402
- [Background] Wereski R, Kimenai DM, Taggart C, Doudesis D, Lee KK, Lowry MTH, Bularga A, Lowe DJ, Fujisawa T, Apple FS, Collinson PO, Anand A, Chapman AR, Mills NL. Cardiac Troponin Thresholds and Kinetics to Differentiate Myocardial Injury and Myocardial Infarction. Circulation. 2021 Aug 17;144(7):528-538. doi: 10.1161/CIRCULATIONAHA.121.054302. Epub 2021 Jun 25. PMID 34167318
- [Background] Greer C, Williams MC, Newby DE, Adamson PD. Role of computed tomography cardiac angiography in acute chest pain syndromes. Heart. 2023 Aug 24;109(18):1350-1356. doi: 10.1136/heartjnl-2022-321360. PMID 36914247
- [Background] Danad I, Fayad ZA, Willemink MJ, Min JK. New Applications of Cardiac Computed Tomography: Dual-Energy, Spectral, and Molecular CT Imaging. JACC Cardiovasc Imaging. 2015 Jun;8(6):710-23. doi: 10.1016/j.jcmg.2015.03.005. PMID 26068288